CLINICAL TRIAL: NCT05538650
Title: Mindfulness-based Social Work and Self-care Study: A Randomised Controlled Trial
Brief Title: RCT: Mindfulness for Social Work and Self-care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Karen McGuigan, Site Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REF167_2122
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Burnout, Professional; Mindfulness; Stress, Psychological; Behaviour
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Behavior | interventions — Self Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Social Work and Self-care (MBSWSC) (Experimental): Participants in the experimental group will participate in the 6 session Mindfulness Based Social Work and Self Care (MBSWSC) programme. MBSWSC is facilitated by two accredited mindfulness practitioners, who are also qualified social workers. Sessions will be supported/supplemented with brief homework activities to help embed mindfulness practice.
  Interventions: Behavioral: Mindfulness-Based Social Work and Self Care (MBSWSC)
- Mindfulness and Self-care (MBSC) (Active Comparator): Participants in the active comparator group will participated in the 3 session Mindfulness and Self-care (MBSC) programme. MBSC is facilitated by two accredited mindfulness practitioners, who are also qualified social workers. Sessions will be supported/supplemented with brief homework activities to help embed mindfulness practice.
  Interventions: Behavioral: Mindfulness-Based Self-Care (MBSC)

INTERVENTIONS:
Behavioral: Mindfulness-Based Social Work and Self Care (MBSWSC) — MBSWSC is a unique mindfulness-based programme for social work and self-care which has been specifically developed for online delivery. The MBSWSC programme is embedded within key cognitive and emotion regulation, and stress coping theory. This programme combines mindfulness practices with psychoeducation with the aim of allowing participants to reduce any negative thinking about the past and future by learning skills that will allow them to focus on the present. It will also focus on how to effectively apply these newly acquired mindfulness skills in social work practice. The programme has been the subject of an initial RCT, which has helped to inform the current programme content and structure. The MBSWSC programme comprises 6x1.5 hour sessions, delivered weekly, over a 6 week period. Homework, in the form of mindfulness practices, is given each week. This will take approximately 20-30 minutes to complete, on 6 out of 7 days, each week.
  Other Names: MBSWSC
  Arms: Mindfulness-based Social Work and Self-care (MBSWSC)
Behavioral: Mindfulness-Based Self-Care (MBSC) — MBSC is a modified, condensed Mindfulness Based Intervention; with a key focus on self-compassion/self-care. Key practices in this condensed programme were chosen for their relevance and utility to social workers. The MBSC programme comprises 3x1 hour sessions delivered over a 6 week period, with one session every two weeks. Homework, in the form of mindfulness practices, is given each week. This will take approximately 20-30 minutes to complete, on 6 out of 7 days, each week.
  Other Names: MBSC
  Arms: Mindfulness and Self-care (MBSC)

SUMMARY:
Social work is a stressful occupation with social workers at high risk of job-related stress and burnout. Mindfulness has been evidenced as a promising approach for improving: recovery from stress; behavioural responses to stress; and resilience.

The Mindfulness-based social work and self-care programme, a bespoke and innovative online mindfulness programme developed for frontline social workers, have been shown to be effective in improving aspects of psychological and general wellbeing among a social work population.

The main aim of the study is to confirm the efficacy of this bespoke, innovative, 6-session Mindfulness Intervention for social workers (MBSWSC) in reducing social worker stress, feelings of burnout, anxiety, low mood and improving well-being. The study will also compare outcomes from the MBSWSC with a briefer, condensed 3 session mindfulness programme (MBSC). The findings of this study will serve to complement and confirm the findings of an initial RCT, but in a post-covid environment.

DETAILED DESCRIPTION:
Background: Social work is a stressful occupation with social workers at high risk of burnout. Existing studies have focused on the impact of working conditions and work-related stress in this population. However, despite this focus stress and burnout among this population remains high, as a result the average working life of social workers considerably shorter than that of counterparts in healthcare.

Interventions to address the impact of job-related stress, and burnout, on frontline social workers have been developed, however there is a lack of evidence on the implementation and effectiveness of these interventions. Robust evidence on effective social work interventions to improve psychosocial outcomes among this population is needed.

Mindfulness is an approach which has been linked to positive outcomes among health and social care professionals, such as improved wellbeing, increased levels of self-compassion, reduced stress and burnout. Self-care or self-compassion has been identified as a promoter of positive health related outcomes among social workers.

However, evidence to support the use of mindfulness interventions among social workers remains scant. There has been a lack of information relating to mindfulness programmes tailored to specific professions; with mindfulness research to date having more of a focus on healthcare or student populations. More information is required on the effectiveness of mindfulness among social workers. An evidence gap also exists around the effectiveness of briefer mindfulness programmes; with recognised programmes such as MBSR and MBCT requiring significant time commitments from participants which may not be suitable for practicing social workers. In light of this evidence it is clear more high quality RCTs are needed to add to the evidence base in this area and to inform future provision for social work.

With this in mind, this study looks to confirm the efficacy of a bespoke, innovative, 6-session Mindfulness Intervention for social workers (MBSWSC); and to explore the mechanisms through which the MBSWSC may mitigate the impact of stress in social work. It also looks to compare the outcomes from the MBSWSC programme with a modified, condensed 3 session mindfulness programme (MBSC) to confirm the impact of briefer mindfulness programmes.

This RCT looks to build on findings of an earlier RCT exploring the effects on MBSWSC. More explicitly, this RCT aims to:

Confirm the efficacy of the MBSWSC programme at improving social worker: - Stress, feelings of burnout, anxiety, low mood and well-being (primary outcomes);

* Mindfulness, attention regulation, acceptance, self-compassion, non-attachment and aversion, worry and rumination (secondary outcomes).
* Explore the mechanisms through which mindfulness may improve outcomes, more specifically the mechanisms through which mindfulness mitigates the effects of stress on burnout.
* Confirm any differences between MBSWSC outcomes and outcomes on the MBSC Methods: A minimum of 70 participants, providing consent to participate in the study will be recruited to the study. On completion of baseline measures, participants will be randomised to either the experimental (MBSWSC) or active control (MBSC) groups. Participants in both groups will complete a range of psychosocial measures at baseline (1 week pre-intervention), post-intervention, and at three month follow-up.

The primary outcome of the study is the efficacy of MBSWSC on social worker stress, feelings of burnout, anxiety, low mood and well-being and secondary outcomes; and the mechanisms through which this occurs.

The secondary outcome of the study is the differences in outcomes for MBSWSC participants and participants on the modified, condensed (briefer) MBSC.

ELIGIBILITY:
Inclusion Criteria:

* Frontline social work practitioner
* Working in Northern Ireland
* Aged 18 years and over

Exclusion Criteria:

* Social workers in strategic social work roles with no contact with clients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Change in Stress measured on the Perceived Stress Scale (PSS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Perceived Stress Scale is a 10-item, reliable and valid, measure of perceived stress. Scores on this scale can range from 0-40, with higher scores indicative of higher levels of stress
Change in Burnout measured on the Maslach Burnout Inventory (MBI) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Maslach Burnout Inventory is a 22-item, reliable and valid measure of work-related burnout. The scale comprises 3 sub scales: burnout, depersonalisation, and personal achievement. The burnout subscale was used in this study. Scores on this sub scale can range from 0-42. Scores of ≤17 on this subscale are indicative of low-level burnout; scores of 18-29 indicate moderate burnout; scores ≥30 indicate high level burnout.
Change in Anxiety measured on the Hospital Anxiety and Depression Scale (HADS-A) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Hospital Anxiety and Depression Scale is a 14-item, reliable and valid measure of anxiety and depression. 7 of the 14 items measure severity of anxiety (HADS-A). Scores on this sub scale can range from 0-21. HADS-A subscale scores of 0-7 are considered normal, whilst scores of 11 or more are classified as moderate to severe
Change in Depression measured on the Hospital Anxiety and Depression Scale (HADS-D) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Hospital Anxiety and Depression Scale is a 14-item reliable and valid measure of anxiety and depression. 7 of the 14 items measure severity of depression (HADS-D). Scores on this sub scale can range from 0-21. HADS-D subscale scores of 0-7 are considered normal, whilst scores of 11 or more are classified as moderate to severe
Change in Wellbeing measured on the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Warwick-Edinburgh Mental Well-being Scale is a 14 item, reliable and valid measure of mental wellbeing. Scores on this scale can range from 14-70. Lower Warwick-Edinburgh Mental Well-being Scale scores are indicative of poorer mental wellbeing

SECONDARY OUTCOMES:
Change in Mindfulness measured by on the Southampton Mindfulness Questionnaire (SMQ) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Southampton Mindfulness Questionnaire is a 16-item reliable and valid measure assessing elements of mindfulness in response to unpleasant thoughts and images. Scores on this scale range from 0-96. Higher scores on the Southampton Mindfulness Questionnaire are indicative of greater levels on mindfulness
Change in Self-compassion measured by on the Self-Compassion Scale (SCS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Self-Compassion Scale is a 12-item reliable and valid measure of self-compassion. Scores on this scale can range from 12-60. Higher mean scores reflect higher levels of self-compassion
Change in Worry measured on the Penn State Worry Questionnaire (PSWQ) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Penn State Worry Questionnaire is a 16-item reliable and valid measure of measure of worry. Scores on this scale can range from 16-80. Higher scores on the Penn State Worry Questionnaire reflect higher levels of pervasive, intense, and uncontrollable worry
Change in Attention Regulation (Decentering) measured on the Experiences Questionnaire - Decentring (EQ-D) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Experiences Questionnaire - Decentring is an 11-item measure of attention regulation/decentering. Scores on this scale range from 11-55. Higher scores on the xperiences Questionnaire - Decentring reflect higher levels of attention regulation
Change in Acceptance measured on the The Philadelphia Mindfulness - Acceptance Subscale (PHLMS-A) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Philadelphia Mindfulness - Acceptance Subscale is a 10-item reliable and valid measure of the mindfulness component of acceptance. Total scores on this sub scale range from 10-50. Lower scores on the Philadelphia Mindfulness - Acceptance subscale reflect higher levels of acceptance
Change in Non-attachment measured by the Southampton Mindfulness Questionnaire Non Attachment subscale (SMQ-LG) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Southampton Mindfulness Questionnaire Non Attachment subscale is a reliable and valid measure of Non-attachment. Scores on this sub scale range from 0-24. Higher scores on this sub scale are indicative of higher levels of non-attachment
Change in Aversion measured by the Southampton Mindfulness Questionnaire Aversion subscale (SMQ-Av) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Southampton Mindfulness Questionnaire Aversion subscale is a reliable and valid measure of Aversion. Scores on this sub scale range from 0-24. Higher scores on this sub scale are indicative of higher levels of aversion
Change in Rumination measured on the Rumination Reflection Questionnaire Rumination subscale (RRQ-R) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Rumination Reflection Questionnaire Rumination subscale is a 12-item measure of engagement in rumination. Scores on this scale range from 12-60. Higher scores on this scale are indicative of greater engagement in rumination

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maddock, Dr, Principal Investigator — University College Dublin
Locations (1):
- Queen's University Belfast, Belfast, Northern Ireland, United Kingdom